CLINICAL TRIAL: NCT02550665
Title: A Multicenter, Randomized, Open-label, Prospective Trial to Evaluate the Safety and Tolerability of Donepezil 23 mg With or Without Intermediate Dose Titration in Patients With Alzheimer's Disease Taking Donepezil Hydrochloride 10 mg
Brief Title: Optimal Dose Escalation Strategy to Successful Achievement of High Dose Donepezil 23mg
Acronym: ODESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A University (Other); Myongji Hospital (Other); Seoul National University Bundang Hospital (Other); Seoul St. Mary's Hospital (Other); Chung-Ang University (Other); Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Jae-Hong Lee, Principal investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHongLee
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- donepezil 15mg titration (Experimental): donepezil 15mg during the first 4 weeks before escalation to 23mg
  Interventions: Drug: donepezil
- donepezil 10mg & 23 mg alternating (Experimental): alternating donepezil 10mg and 23mg during the first 4 weeks before escalation to 23mg
  Interventions: Drug: donepezil
- no titration of donepezil (Active Comparator): no titration and direct escalation to 23mg donepezil
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: donepezil — using different titration method for the first 4 weeks, and after the 4 weeks, 23mg/day orally
  Other Names: aricept

SUMMARY:
This study evaluates the side effects of dose escalation in the treatment of donepezil 23mg for patients with Alzheimer's disease. Investigators randomly divide participants into three groups according to the dose escalation method; no titration, 15mg of donepezil for a month before escalation to 23mg, and alternating of 10mg and 23mg for a month before escalation to 23mg.

DETAILED DESCRIPTION:
High dose of donepezil is currently prescribed for patients with Alzheimer's disease who showed poor response in lower dose, however the side effect profiles according to dose titration method were not clarified yet. This study aims to confirm which titration method would show better safeties and tolerabilities in the high dose donepezil treatment. Investigators include patients with moderate to severe dementia who were diagnosed as probable Alzheimer's disease and treated with donepezil 10mg at least 3 months before the study. The study duration is for 12 weeks and the titration duration is the first 4 weeks of the study. Investigators evaluate the side effects profiles and vital signs at every 4 weeks and measure blood laboratory tests at screening and the last visit.

ELIGIBILITY:
Inclusion Criteria:

* dementia according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria
* probable Alzheimer's disease dementia according to National Institute on Aging-Alzheimer's Association (NIAAA) criteria
* Mini-Mental State Examination (MMSE) score of 20 or less
* General Deterioration Scale (GDS) score of 4 or more / Clinical Dementia Rating (CDR) score of 2 or more
* stable dose of 10mg donepezil at least 3 months before screening
* caregiver who can come together at every visit and give informations about side effects profiles should exist
* patients and caregivers accepted the study

Exclusion Criteria:

* patients receiving other concomitant acetylcholinesterase inhibitor
* uncontrolled psychiatric disorders
* drug overuse or alcohol abuse history within 5 years
* significant uncontrolled or active medical conditions
* uncontrolled epilepsy
* patients who cannot come at scheduled visits

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | Change from baseline at 4 week
  adverse events (nausea, vomiting, diarrhea, anorexia, abdominal pain, headache and other unpredicted adverse events)are asked and assessed using 3 grade scale (mild, moderate, severe)

SECONDARY OUTCOMES:
blood WBC | 12 week
  if WBC count is below 4000/uL or above 10000/uL, abnormal
blood BUN | 12 week
  if BUN level is above 30 mg/dL, abnormal
blood Creatinine | 12 week
  if creatinine level is above 1.4 mg/dL, abnormal
blood sodium | 12 week
  if sodium level is below 135mmol/L or above 145mmol/L, abnormal
blood potassium | 12 week
  if potassium level is below 3.5mmol/L or above 5.1mmol/L, abnormal
blood AST/ALT | 12 week
  if AST or ALT level is above 50 IU/L, abnormal
weight loss | 4 week, 8 week, 12 week
  if the weight is decreased over 5% of body weight at screening visit, then weight loss
drug compliance (counting of residual drug) | 4 week, 8 week, 12 week
  if the (number of prescribed drugs - number of residual drugs)/ number of prescribed drugs is below 80%, then consider as low compliance, if compliance is between 80-100% then consider as good compliance
heart rate on Electrocardiography (ECG) | 12 week
  checking whether heart rate on ECG is normal because donepezil can cause bradycardia; if the heart rate is decreased below 50, then write down as bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong YJ, Han HJ, Youn YC, Park KW, Yang DW, Kim S, Kim HJ, Kim HJ, Lee Y, Kwon M, Lee JH; ODESA study (Optimal Dose Escalation Strategy to Successful Achievement of High Dose Donepezil 23 mg). Effects of Body Weight on the Safety of High-Dose Donepezil in Alzheimer's Disease: Post hoc Analysis of a Multicenter, Randomized, Open-Label, Parallel Design, Three-Arm Clinical Trial. Dement Geriatr Cogn Disord. 2021;50(3):289-295. doi: 10.1159/000518470. Epub 2021 Sep 10. PMID 34518459
- [Derived] Hong YJ, Han HJ, Youn YC, Park KW, Yang DW, Kim S, Kim HJ, Kim JE, Lee JH; ODESA study (Optimal Dose Escalation Strategy to Successful Achievement of High Dose Donepezil 23 mg). Safety and tolerability of donepezil 23 mg with or without intermediate dose titration in patients with Alzheimer's disease taking donepezil 10 mg: a multicenter, randomized, open-label, parallel-design, three-arm, prospective trial. Alzheimers Res Ther. 2019 May 1;11(1):37. doi: 10.1186/s13195-019-0492-1. PMID 31039806